CLINICAL TRIAL: NCT00163709
Title: A Randomised Trial of BNP Testing in Patients With Shortness of Breath in the Emergency Department to Improve Patient Outcome
Brief Title: BNP Testing in Patients With SOB on Presentation to ED
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Collaborators: The Alfred (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 116/05; Heart Foundation Grant
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2006-10-04 (Estimated); Status verified 2005-05

CONDITIONS: Heart Failure, Congestive
Keywords: Atrial natriuretic factor.; Biochemistry.; Cardiac failure.; Randomised trials.; Hormones.; Systolic heart failure.; Diastolic heart failure.; Ischaemic cardiomyopathy.; Ventricular hypertrophy.; AMI
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic; Heart Failure, Diastolic

INTERVENTIONS:
Procedure: BNP test

SUMMARY:
A trial to examine whether a new heart failure blood test can improve the outcome of patients presenting to the Emergency Department with shortness of breath.

We hypothesise that a BNP test performed in real-time in patients presenting to the Emergency Department with shortness of breath will help identify additional patients with CHF and consequently to change practice and allow more patients to recieve correct treatment earlier.

DETAILED DESCRIPTION:
In recent years new tests to diagnose heart failure have become available. We are evaluating a new test called B-type natriuretic peptide(BNP)in patients presenting to the Emergency Department with shortness of breath. Patients are randomised into whether they will receive the new test or not. In the patient group where the test is positive, standardised approach that will optimise heart failure treatment will be introduced. We hypothesise that with this approach we will improve the clinical care of patients who present to the Emergency Department with shortness of breath. Measures of outcomes will be the accuracy of diagnosis 2 hours after presentation, 30 day mortality, hospital and ICU admission rates and quality of life at 30days.

We plan to investigate 600 consecutive patient presenting to the to the Emergency Department with shortness of breath that are over 40 years old and present with an emergency department triage category of 3 or higher. Patients presenting with a traumatic cause of dyspnea, patients with severe renal disease, patients with cardiogenic shock and patients who have early transfer to another hospital(within 24 hrs) will be excluded.

ELIGIBILITY:
Inclusion Criteria:

We plan to include all patients presenting to the ED with shortness of breath that are over 40 years old and present with an emergency department triage category of 3 or higher.

Exclusion Criteria:

Patients presenting with a traumatic cause of dyspnea, patients with severe renal disease (serum creatinine level of more than 250 micro mmol/L, patients with cardiogenic shock, and patients who have an early transfer to another hospital (within 24 hrs) will be excluded.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2005-08

PRIMARY OUTCOMES:
Allow more accurate diagnosis of heart failure.
Cause a change of management.
Benefit some patients presenting with shortness fo breath more than others.
Increse the use of early Continuous Positive Airway Pressure (CPAP) ventilation, nitrates, loop diuretics and ACE inhibitors.
Decrease hospital stay.
Decrease hospital admission rate.
Decrease the number of endotracheal intubations.
Decrease 30-day mortality.

SECONDARY OUTCOMES:
Improve long term outcomes in the Australian setting.
Improve cost effectiveness in the Australian setting.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Schneider, MBBS, Principal Investigator — Head, Pathology Department
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Lokuge A, Lam L, Cameron P, Krum H, de Villiers S, Bystrzycki A, Naughton MT, Eccleston D, Flannery G, Federman J, Schneider HG. B-type natriuretic peptide testing and the accuracy of heart failure diagnosis in the emergency department. Circ Heart Fail. 2010 Jan;3(1):104-10. doi: 10.1161/CIRCHEARTFAILURE.109.869438. Epub 2009 Nov 20. PMID 19933409
- [Derived] Schneider HG, Lam L, Lokuge A, Krum H, Naughton MT, De Villiers Smit P, Bystrzycki A, Eccleston D, Federman J, Flannery G, Cameron P. B-type natriuretic peptide testing, clinical outcomes, and health services use in emergency department patients with dyspnea: a randomized trial. Ann Intern Med. 2009 Mar 17;150(6):365-71. doi: 10.7326/0003-4819-150-6-200903170-00004. PMID 19293069